CLINICAL TRIAL: NCT02710955
Title: Study on the Tolerance and Efficacy of a New Anti-regurgitation Formula (PC-2016-01)
Brief Title: SWAN: Study on the Tolerance and Efficacy of a New Anti-regurgitation Formula (PC-2016-01)
Acronym: SWAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01-SWAN
Record Dates: First submitted 2016-03-08; First posted 2016-03-17 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-05

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thickened infant formula (Experimental)
  Interventions: Dietary Supplement: Thickened infant formula

INTERVENTIONS:
Dietary Supplement: Thickened infant formula

SUMMARY:
The aim of this study is to evaluate the efficacy of a new thickened formula on regurgitation

ELIGIBILITY:
Inclusion Criteria:

* Infants :

  * Aged ≤ 5 months old
  * fully formula fed
  * with at least 5 episodes of regurgitation per day, for at least a week

Exclusion Criteria:

* Breast fed infants
* Infants presenting symptoms of a complicated gastroesophageal reflux
* Infants presenting intestinal disorders

Ages: 1 Week to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-04-01; Primary Completion 2017-01-21 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Number of episodes of regurgitation per day | 14 days

SECONDARY OUTCOMES:
Regurgitation score assessed through Vandenplas score | 14 and 90 days
Stools frequency over 72h | 14 and 90 days
Stools consistency assessed through Bristol Stool form Scale | 14 and 90 days
Weight expressed in z scores according to the WHO Child Growth Standards | 90 days
Height expressed in z scores according to the WHO Child Growth Standards | 90 days
BMI expressed in z scores according to the WHO Child Growth Standards | 90 days
Head circumference expressed in z scores according to the WHO Child Growth Standards | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yvan Vandenplas, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis, Brussels, Belgium